CLINICAL TRIAL: NCT05108545
Title: A Multicenter, Open-label, Phase Ⅲ Study to Evaluate the Efficacy and Safety of Amphotericin B Liposome for Injection in Patients With Persistent Febrile Neutropenia
Brief Title: A Study of Amphotericin B Liposome for Injection in Patients With Persistent Neutropenia and Fever
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC1507-CSP-001
Record Dates: First submitted 2021-09-30; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-09

CONDITIONS: Neutropenia and Fever
MeSH Terms: conditions — Neutropenia; Fever | interventions — Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amphotericin B liposomes (Experimental): Patients with suspected fungal neutropenia and fever will receive amphotericin B liposome 3 mg/kg intravenously. Treatment will be continued until the ANC≥500 /mm^3 (0.5×10^9 /L) for more than 72 hrs in terms of patients without evidence of baseline fungal infection and breakthrough fungal infection; or treatment will be continued according to investigator's judgement with a duration ranging from 14 days to 12 weeks in terms of patients with evidence of baseline fungal infection and breakthrough fungal infection.
  Interventions: Drug: Amphotericin B liposomes

INTERVENTIONS:
Drug: Amphotericin B liposomes — Amphotericin B liposomes for injection, 3 mg/kg, qd, IV

SUMMARY:
This is a multicenter, open-label, single-arm, phase III study to evaluate the safety and efficacy of Amphotericin B liposomes in patients with persistent neutropenia and fever.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase III study to evaluate the safety and efficacy of Amphotericin B liposomes in patients with persistent neutropenia and fever. About 93 patients will be recruited in this study. The patients will receive Amphotericin B liposomes intravenous infusion at a dose of 3 mg/kg over 2 hours once daily (qd) for a maximum of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 ~ 75 years (inclusive), no gender limitation.
2. Patients with neutrophilic deficiency after solid tumor chemotherapy, hematological tumor chemotherapy, hematopoietic stem cell transplantation, etc. (absolute neutrophil count (ANC) in peripheral blood <500 /mm^3 (0.5×10^9 /L) for at least 72 hours at screening).
3. Persistent or recurrent fever (oral temperature ≥38℃ or axillary temperature ≥37.7℃ within 24 hours prior to randomization) after at least 72 hours on broad-spectrum antibiotics, and considering fever to be associated with suspected fungal infection.
4. Female patients must meet one of the following conditions:

   1. Menopausal patients, menopause at least 1 year;
   2. Patients of childbearing age: Negative for blood/urine pregnancy test before enrollment; agree to take a guaranteed, effective contraception during the study and within 4 weeks after the study.
5. Male patients and their partners must use effective contraception throughout the study period and up to 4 weeks after leaving the study.
6. Patients fully understand and voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

1. History of allergy to liposomes or amphotericin B.
2. Received systemic treatment of amphotericin B or amphotericin B-containing formulation within 10 days prior to enrollment.
3. Liposome used within 1 month before the signing informed consent.
4. Confirmed or clinically diagnosed invasive fungal infection or known uncontrolled bacteremia or sepsis at screening.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≥3;
6. Abnormal liver function, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≥5 × the upper limit of normal (ULN), or ALT/AST ≥3 × ULN with total bilirubin ≥1.5 × ULN, or total bilirubin ≥3 × ULN.
7. Serum creatinine > 2 × ULN.
8. Serum potassium concentration ≤3.0 mmol/L prior to the first administration, or serum potassium concentration ≤the lower limit of normal value (LLN) in patients undergoing digitalization.
9. 12-lead ECG presenting II or III degree atrioventricular block, long QT syndrome or corrected QT interval>480 ms in the absence of a pacemaker.
10. Cardiac function grade III/IV (NYHA).
11. Tachyarrhythmia requiring intervention and a history of high-risk coronary heart disease such as unstable angina and acute coronary syndrome.
12. Human immunodeficiency virus (HIV) antibody or treponema pallidum specific antibody (TPHA) positive; active tuberculosis on CT of chest (to be determined by investigator).
13. Pregnant or lactating female.
14. A history of drug abuse (non-medical use of narcotic drugs or psychotropic substances) or drug dependence (narcotics, stimulants and psychotropic substances, etc.) within 2 years.
15. Plan to use prohibited drugs during the study period.
16. Enrolled in any other clinical trials of drugs or medical devices within 3 months prior to screening.
17. Life expectancy < 2 months;
18. Not suitable for this study as decided by the investigator due to other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall success rate | From the initiation of the third dose to 7 days after the last dose
  A successful outcome is defined as fulfilling all components of a prespecified 5-part composite endpoint.

SECONDARY OUTCOMES:
Percentage of patients without new fungal infections from the initiation of the first dose to 7 days after the last dose | From the initiation of the third dose to 7 days after the last dose
  Percentage of patients without new fungal infections
Percentage of patients survived from the initiation of the first dose to 7 days after the last dose | From the initiation of the third dose to 7 days after the last dose
  Percentage of patients survived
Percentage of patients without discontinuation of study drug due to side effects or lack of efficacy during the treatment period | From the initiation of the third dose to 7 days after the last dose
  Percentage of patients without discontinuation of study drug due to side effects or lack of efficacy
Percentage of patients experienced fever reduction during neutropenia after initiation of treatment | From the initiation of the third dose to 7 days after the last dose
  Percentage of patients experienced fever reduction during neutropenia
Percentage of patients with complete or partial remission of confirmed or clinically diagnosed IFD (baseline fungal infection) at the end of treatment | From the initiation of the third dose to 7 days after the last dose
  Percentage of patients with complete or partial remission of confirmed or clinically diagnosed Invasive fungal disease (baseline fungal infection)
Adverse events | From the screening period to 14 days after the last dose
  Adverse events
Pharmacokinetic profile of amphotericin B | Pre-dose and multiple timepoints up to 4 hours of the last dose
  Pharmacokinetic profile of amphotericin B, Such as "Peak Plasma Concentration (Cmax)"
Pharmacokinetic profile of amphotericin B | Pre-dose and multiple timepoints up to 4 hours of the last dosePharmacokinetic profile of amphotericin B, Such as "Area under the plasma concentration versus time curve (AUC)"